CLINICAL TRIAL: NCT01555801
Title: Efficacy Study of Endoscopic Ultrasound Combining With Submucosal Saline Injection for Pretreatment Staging of T1a and T1b in Patients With Early Esophageal Cancer
Brief Title: Endoscopic Ultrasound Plus Submucosal Injection for Early Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 112273; 1122 (Registry Identifier: Jian-jun Li)
Record Dates: First submitted 2012-02-29; First posted 2012-03-15 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; early cancer; ultrasonography (EUS); stage
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Endosonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Submucosal injection combining with EUS (Experimental): The enrolled patients will be accepted submucosal injection of saline,then ultrasonography will performed(EUS+SIS group).So,stages of EUS in these early esophageal cancer will be recorded and compared with the pathological stages afer endoscopic mucosal resection(EMR) or endoscopic submucosal dissection(ESD) or esophagectomy.
  Interventions: Device: submucosal injection needle ; EUS
- ordinary endosonography(EUS) (Placebo Comparator): The enrolled patients will accept ordinary ultrasonography .So,stages of EUS in these early esophageal cancer will be recorded and compared with the pathological stages afer endoscopic mucosal resection(EMR) , endoscopic submucosal dissection(ESD) or esophagectomy.
  Interventions: Device: ordinary endosonography(EUS)

INTERVENTIONS:
Device: submucosal injection needle ; EUS — The patients will accepted submucosal injection of 5ml saline followed by ordinary endosonography(EUS) before surgery or endoscopic dissection.
  Other Names: submucosal injection needle:Olympus,NM-20K-0423;; EUS:Olympus,UM2000
  Arms: Submucosal injection combining with EUS
Device: ordinary endosonography(EUS) — These patients will be accepted ordinary EUS followed by surgery or endoscopic dissection.
  Other Names: EUS:Olympus,UM2000
  Arms: ordinary endosonography(EUS)

SUMMARY:
Preoperative accurately staging T1a or T1b in early esophageal cancer is vital for the choices of treatment. At present, the main diagnostic method for early esophageal cancer is endoscopic ultrasound (EUS). However, the accuracy of EUS alone is poor. Thus, it is necessary to improve endoscopic ultrasound examination methods. This project is concerning on the efficacy of EUS combining with submucosal injection of saline for staging T1a and T1b-esophageal cancer. Patients and methods: 80 cases of pathological confirmed early esophageal cancer were randomly divided into two groups: endoscopic ultrasonography group (EUS group) and EUS combining with submucosal injecting saline group (EUS+SIS group). All the cases will be performance by endoscopic or surgical resection; postoperative pathologic diagnosis will be obtained involving echo, depth, margin and other features. The EUS results of two groups of patients will be compared with pathologic results. From comparison, the efficacy and accuracy of EUS+SIS for staging T1a and T1b in esophageal cancer patients will be validated. Through this study, the investigators may develop a routine diagnostic and accurately staging method for early esophageal cancer patients.

DETAILED DESCRIPTION:
Someone whom may concern our IPD are available to the PI, Jian-jun Li M.D. or at lijj@sysucc.org.cn

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, no gender limited;
* Patients with esophageal squamous cell carcinoma who be confirmed by ordinary endoscopy and pathologic biopsy;
* Patients who agree to accept endoscopic resection or surgical excision of the lesion in esophagus;
* patients with normal cardio-pulmonary function and normal coagulative function,are predicted to be tolerated anesthesia and surgery;
* patients who understand test purpose, volunteer to join these study and sign the consent inform.

Exclusion Criteria:

* Patients with stages of T2, T3, or T4 displayed by EUS;
* Patients who can't tolerate endoscopy and surgical treatment for various reasons;
* Patients who have distant metastasis, or multiple source of malignant tumors;
* Patients with blood coagulative disorder;
* Patients don't accept the endoscopic examination or surgical treatment;
* Patients with poor compliancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Participants will be followed for the duration of hospital stay in order to accept endosopic or surgical resection , an expected average of 10 days
  The stages judged from submucosal injection plus EUS or ordinary EUS will be compared with the pathological results after endoscopic or surgical resection.So the sensitivity,specificity,positive predictive value,negative predictive value and diagnostic accuracy of either submucosal injection plus EUS or ordinary EUS for early esophageal cancer will be measured respectivly.
Specificity | Participants will be followed for the duration of hospital stay in order to accept endosopic or surgical resection , an expected average of 10 days
  As well as sensitivity described above.
Diagnostic accuracy | Participants will be followed for the duration of hospital stay in order to accept endosopic or surgical resection , an expected average of 10 days
  As well as sensitivity described above.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- cancer center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] He LJ, Xie C, Wang ZX, Li Y, Xiao YT, Gao XY, Shan HB, Luo LN, Chen LM, Luo GY, Yang P, Zeng SC, Xu GL, Li JJ. Submucosal Saline Injection Followed by Endoscopic Ultrasound versus Endoscopic Ultrasound Only for Distinguishing between T1a and T1b Esophageal Cancer. Clin Cancer Res. 2020 Jan 15;26(2):384-390. doi: 10.1158/1078-0432.CCR-19-1722. Epub 2019 Oct 15. PMID 31615934